CLINICAL TRIAL: NCT04357899
Title: Stroke Research Consortium in Northern Bavaria - STAMINA, a Multicenter Longitudinal Cohort Study on Ischemic Stroke Treatment
Brief Title: Stroke Research Consortium in Northern Bavaria (STAMINA)
Acronym: STAMINA
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 33_20B
Record Dates: First submitted 2020-04-16; First posted 2020-04-22 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2021-04

CONDITIONS: Ischemic Stroke
Keywords: Thrombolysis; Mechanical thrombectomy; Endovascular procedure; Stroke; Cerebrovascular Disorders; Brain Diseases; Brain Ischemia; Cerebral Infarction; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Tissue Plasminogen Activator; Fibrinolytic Agents; Fibrin Modulating Agents
MeSH Terms: conditions — Ischemic Stroke; Stroke; Cerebrovascular Disorders; Brain Diseases; Brain Ischemia; Cerebral Infarction; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Thrombolytic Therapy; Fibrinolytic Agents; Multimodal Imaging; Secondary Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: thrombolysis therapy
  Other Names: thrombolytic drugs
Procedure: endovascular therapy
Procedure: decompressive surgery
Diagnostic Test: multimodal imaging in acute ischemic stroke
Procedure: transfer of acute stroke patients to tertiary stroke centers
Drug: initiation of antiplatelets, oral anticoagulation and lipid lowering drugs for secondary prevention
  Other Names: antithrombotic oder lipid lowering drugs

SUMMARY:
Each year, approximately 15 million people suffer a stroke worldwide of which 80% are due to ischemic cerebral infarction. Based on the results of randomized controlled trials, treatment options and patient outcomes in acute ischemic stroke have dramatically improved in recent years. However, these advances in thrombolysis and endovascular therapy need to be established outside controlled trials to optimize stroke management, treatment procedures, patient selection and inter-hospital transfer in clinical practice. This multicenter longitudinal cohort study is based on a large stroke care network in Northern Bavaria, Germany (region of more than 3.5 million inhabitants) to evaluate and improve treatment in ischemic stroke.

DETAILED DESCRIPTION:
Methods: This multicenter longitudinal cohort study will include ischemic stroke patients treated within a telemedical stroke care network and patients transferred to tertiary stroke centers for treatment procedures from hospitals outside the telemedical network. Individual patient data are available from two tertiary stroke centers and 24 primary and secondary stroke facilities in Northern Bavaria, Germany. Patients with ischemic stroke transferred to the tertiary stroke centers for treatment procedures - i.e. endovascular therapy or thrombolysis in stroke with an unknown time of onset - and all stroke patients with either large vessel occlusion (LVO) and/or thrombolysis therapy admitted to the University Hospital Erlangen will be integrated from institutional prospective stroke registries. Consecutive patients admitted between January 2006 and December 2019 will be included, an estimated total number of more than 3000 ischemic stroke patients - approximately 1000 patients with LVO receiving endovascular therapy, 1000 patients with LVO not receiving endovascular therapy and 1000 patients without LVO receiving thrombolysis therapy.

Demographic and clinical data including medical history, medication and laboratory results will be obtained by review of medical charts, institutional databases or prospective registries, supplemented by structured interviews on follow-up information or by review of all available medical records. In detail the following parameters will be evaluated: prior medical history (e.g. comorbidities, premorbid functional status, medication), admission status (e.g. NIHSS, GCS, body temperature, arterial blood pressure), cerebral imaging parameters (e.g. Alberta Stroke Program Early CT score [ASPECTS], perfusion volumes, mismatch and collateral status on admission imaging, final infarct volume on follow-up imaging), treatment procedures (e.g. intravenous thrombolysis, endovascular therapy, decompressive surgery), time intervals (e.g. symptom onset or last seen normal until admission, imaging, thrombolysis, groin puncture, recanalization), complications (e.g. hemorrhagic transformation, arterial dissection, distant ischemic stroke), laboratory parameters, clinical and diagnostic follow-up (e.g. neurological status, blood pressure, vascular ultrasound), stroke etiology, secondary prevention (e.g. lipid lowering medication, antiplatelet therapy, anticoagulation) and clinical outcomes (e.g. mortality, modified Rankin Scale).

Ethics Approval: The study was approved by the Institutional Review Board of the Friedrich-Alexander-Universität Erlangen-Nürnberg.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms consistent with the diagnosis of an acute ischemic stroke
* Presence of large vessel occlusion (as evidenced by CTA, MRA or DSA) and/or intravenous thrombolysis therapy applied

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke patients treated within a stroke care network in Northern Bavaria, Germany.
Sampling Method: Probability Sample
Enrollment: 3769 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Functional Outcome (modified Rankin Scale 0-6) | at day 90
  The Distribution of Scores on the modified Rankin Scale (mRS)
Functional Independence (modified Rankin Scale 0-2) | at day 90
  Proportion of participants with functional independence (mRS 0-2)
Favorable Outcome (modified Rankin Scale 0-1) | at day 90
  Proportion of participants with favorable outcome (mRS 0-1)
Infarct volume | at day 5 (±2)
  Infarct volume on CT or diffusion-weighted MRI
Lesion growth volume | at day 5 (±2)
  Lesion growth volume between ischemic core on baseline imaging and infarkt volume
Intracranial hemorrhage | at 24 (±6) hours
  Rate of intracranial hemorrhage defined according to different criteria (ECASS II, SITS-MOST, NINDS or Parenchymal hemorrhage Type 2) on the 24 hour scan
Recanalization Rates | at 24 (±6) hours
  Recanalization of the primary arterial occlusive lesion (based on ultrasound, clinical and radiological assessment) at 24-hours

SECONDARY OUTCOMES:
Mortality | at 90 days
  All cause mortality rate
Procedure time | procedure
  Time from groin puncture to first recanalization
Door-to-groin puncture time | until 24 hours after admission to the tertiary stroke center or until hospital discharge, whichever came first
  Time from arrival at the tertiary stroke center to groin puncture
Door-to-needle time | until 24 hours after admission to the tertiary stroke center or until hospital discharge, whichever came first
  Time from hospital arrival to IVT administration
Symptom-to-door time | until 24 hours after admission to the tertiary stroke center or until hospital discharge, whichever came first
  Time from symptom onset to arrival at the first hospital
Interhospital transfer time | until 24 hours after admission to the tertiary stroke center or until hospital discharge, whichever came first
  Time from arrival at the first hospital to arrival at the tertiary stroke center

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schwab, Principal Investigator — Friedrich-Alexander-Universität (FAU) Erlangen-Nürnberg, Department of Neurology, Germany; Arnd Dörfler, Principal Investigator — Friedrich-Alexander-Universität (FAU) Erlangen-Nürnberg, Department of Neuroradiology, Germany; Bernd Kallmünzer, Principal Investigator — Friedrich-Alexander-Universität (FAU) Erlangen-Nürnberg, Department of Neurology, Germany; Tobias Engelhorn, Principal Investigator — Friedrich-Alexander-Universität (FAU) Erlangen-Nürnberg, Department of Neuroradiology, Germany
Locations (2):
- Germany (2):
  - Institut für Neuroradiologie, Universitätsklinikum Erlangen, Erlangen
  - Neurologische Klinik, Universitätsklinikum Erlangen, Erlangen

IPD SHARING:
Plan to Share IPD: Undecided
Because of local ethics committees restrictions the final decision upon release of the raw data has not been made.

REFERENCES:
- [Derived] Macha K, Sembill JA, Muehlen I, Engelhorn T, Doerfler A, Schwab S, Kallmunzer B. IV Thrombolysis for Acute Ischemic Stroke with Unknown Onset in Patients on Oral Anticoagulation. Cerebrovasc Dis. 2025;54(4):499-507. doi: 10.1159/000540552. Epub 2024 Aug 23. PMID 39182487
- [Derived] Sembill JA, Sprugel MI, Haupenthal D, Kremer S, Knott M, Muhlen I, Kallmunzer B, Kuramatsu JB. Endovascular thrombectomy in patients with anterior circulation stroke: an emulated real-world comparison. Neurol Res Pract. 2024 Jul 25;6(1):37. doi: 10.1186/s42466-024-00331-6. PMID 39049127